CLINICAL TRIAL: NCT04746053
Title: Study of Ovarian Function and Gynecological Profile of Patients Carrying a Pathogenic Variant of the HNF1B Gene (GYN-HNF1)
Brief Title: Ovarian Function and Gynecological Profile of Patients Carrying a Pathogenic Variant of the HNF1B Gene (GYN-HNF1)
Acronym: GYN-HNF1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/20/0124; 2020-A02800-39 (Other: ID-RCB)
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Genital Diseases, Female
Keywords: gene HNF1b mutation; ovarian function; genital malformations
MeSH Terms: conditions — Genital Diseases, Female | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient with a mutation in the HNF1B gene (Other): Patient with a mutation in the HNF1B gene and which are followed in the reference centers
  Interventions: Other: Pelvic ultrasound; Biological: blood sample

INTERVENTIONS:
Other: Pelvic ultrasound — Pelvic or vaginal ultrasound
Biological: blood sample — blood sample (5ml)

SUMMARY:
The main objective of this study is to study the ovarian function of patients with hepatocyte nuclear factor-1beta (HNF1B) abnormality, followed in the reference centers of Toulouse and Paris University Hospitals. The secondary objectives are to know the gynecological profile of these patients.

A dosage of anti-mullerian hormone (AMH) will be added to the usual balance, whatever the phase of the cycle and a pelvic ultrasound will be performed by the same operator by center. Patients will be received in a dedicated consultation to complete a questionnaire on gynecological and obstetric history, as well as their personal and family history. There will be no gynecological examination during this consultation.

DETAILED DESCRIPTION:
HNF1B mutations can be responsible for genital malformations associated with renal development abnormalities. HNF1b is also a candidate gene involved in the development of the renal tract and the Mullerian system but there is no data in the literature regarding the ovarian function and clinical gynecological profile of these patients.

The main objective of this study is to study the ovarian function of patients with HNF1B abnormality, followed in the reference centers of Toulouse and Paris University Hospitals. The secondary objectives are to know the gynecological profile of these patients.

A dosage of AMH will be added to the usual balance, whatever the phase of the cycle and a pelvic ultrasound will be performed. Patients will be received in a dedicated consultation to complete a questionnaire on gynecological and obstetric history, as well as their personal and family history. There will be no gynecological examination during this consultation.

ELIGIBILITY:
Inclusion Criteria:

* Girls from 12 years of age carrying a pathogenic variant of the HNF1 B gene and monitored in the reference center for rare renal diseases
* Person affiliated or beneficiary of a social security scheme.
* Free, informed and written consent signed by the participant or her legal representative if a minor patient and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Woman unable to answer
* Pregnant or breastfeeding woman
* Refusal of participation by the patient or her legal representative
* Person under a protection system for adults (such as safeguard of justice, guardianship or curatorship)
* History of chemotherapy, radiotherapy, brachytherapy
* History of ovarian endometrium

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
serum level of Antimullerian Hormone levels | day 1
  serum level of antimullerian hormone levels in ng/mL

SECONDARY OUTCOMES:
ultrasound result | day 1
  ultrasound (pelvic or vaginal) will allow the team to look at whether or not there is a genital defect and the type of defect.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine PIENKOWSKI, MD, Principal Investigator — University Hospital, Toulouse
Locations (3):
- France (3):
  - Pitié Salpêtrière Hospital -, Paris
  - Necker Hospital, Paris
  - Toulouse University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edghill EL, Bingham C, Ellard S, Hattersley AT. Mutations in hepatocyte nuclear factor-1beta and their related phenotypes. J Med Genet. 2006 Jan;43(1):84-90. doi: 10.1136/jmg.2005.032854. Epub 2005 Jun 1. PMID 15930087
- [Background] Lindner TH, Njolstad PR, Horikawa Y, Bostad L, Bell GI, Sovik O. A novel syndrome of diabetes mellitus, renal dysfunction and genital malformation associated with a partial deletion of the pseudo-POU domain of hepatocyte nuclear factor-1beta. Hum Mol Genet. 1999 Oct;8(11):2001-8. doi: 10.1093/hmg/8.11.2001. PMID 10484768
- [Background] Oram RA, Edghill EL, Blackman J, Taylor MJ, Kay T, Flanagan SE, Ismail-Pratt I, Creighton SM, Ellard S, Hattersley AT, Bingham C. Mutations in the hepatocyte nuclear factor-1beta (HNF1B) gene are common with combined uterine and renal malformations but are not found with isolated uterine malformations. Am J Obstet Gynecol. 2010 Oct;203(4):364.e1-5. doi: 10.1016/j.ajog.2010.05.022. Epub 2010 Jul 15. PMID 20633866